CLINICAL TRIAL: NCT01655394
Title: Change of Nerve Conduction Properties in IVIg Dependent Neuropathies
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Helmar Lehmann, PD Dr. med. H. Lehmann, University of Cologne
Other Study IDs: 01607831337
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Guillain-Barre Syndrome; CIDP; Multifocal Motor Neuropathy
MeSH Terms: conditions — Guillain-Barre Syndrome; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
IVIg exert a variety of different immunomodulatory effects and several mechanism of action have been proposed for IVIg. In this study the role of IVIg on short term nerve conduction in patients with immune-mediated neuropathies will be explored.

DETAILED DESCRIPTION:
IVIg exert a variety of different immunomodulatory effects and several mechanism of action have been proposed for IVIg. In this study the role of IVIg on short term nerve conduction in patients with immune-mediated neuropathies will be explored

ELIGIBILITY:
Inclusion Criteria:

* immune neuropathy
* age above 18 y
* IVIg treatment

exclusion:

* no IVIg treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with immune neuropathies
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Helmar C. Lehmann, PD Dr. med., Principal Investigator — PI
Locations (1):
- University of Cologne, Cologne, Germany